CLINICAL TRIAL: NCT02297464
Title: Eggs as Part of a Healthy Breakfast: Lack of Association With Heart Disease Risk
Brief Title: Eggs as Part of a Healthy Breakfast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Maria Luz Fernandez, Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: H14-032
Record Dates: First submitted 2014-11-13; First posted 2014-11-21 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Cardiovascular Diseases
Keywords: Risk
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Breakfast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eggs - 2 per day for breakfast (Experimental): Participants will consume 2 eggs per day for breakfast for 4 weeks of the study.
  Interventions: Other: Eggs - 2 per day for breakfast; Other: 1 packet of oatmeal per day
- Oatmeal - 1 packet per day for breakfast (Experimental): Participants will consume 1 packet of oatmeal per day for breakfast for 4 weeks of the study.
  Interventions: Other: Eggs - 2 per day for breakfast; Other: 1 packet of oatmeal per day

INTERVENTIONS:
Other: Eggs - 2 per day for breakfast — 11-week crossover study in which participants consumed 2 eggs or 1 packet of oatmeal per day daily for 4 weeks, separated by a 3-week washout period.
Other: 1 packet of oatmeal per day — 11-week crossover study in which participants consumed 2 eggs or 1 packet of oatmeal per day daily for 4 weeks, separated by a 3-week washout period.

SUMMARY:
Contrary to popular belief, previous studies have demonstrated beneficial effects of whole egg consumption in modifying biomarkers indicative of a greater risk of coronary heart disease (CHD), chronic inflammation, and insulin resistance. The following study is designed to conduct a comprehensive evaluation of consuming an egg-based breakfast compared to an oatmeal-based breakfast on lipid biomarkers, oxidative stress, inflammation, insulin sensitivity, and satiety in young, healthy men and women. The investigators hypothesize that the consumption of 2 eggs per day will not negatively impact plasma lipids in a young, healthy population.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-30, willing to consume eggs and oatmeal daily, proficient in English, and with a healthy lipid profile.

Exclusion Criteria:

* Currently have liver disease, renal disease, diabetes, cancer, history of stroke or heart disease
* Currently taking glucose lowering drugs or supplements
* Plasma triglycerides >500 mg/dL, glucose >126, total cholesterol >240
* Pregnant, lactating, or have endocrine or metabolic disorders
* BMI ≥ 30
* Blood pressure > 140/90 (average of 3 readings)
* Allergies to eggs
* Celiac disease or gluten sensitivity

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Spectrophotometry, NMR and ELISA will assess plasma lipids. | 1 year

SECONDARY OUTCOMES:
Visual analog scales (VAS) and ELISA assays will assess satiety. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States